CLINICAL TRIAL: NCT01651611
Title: Health Advocates as a Vehicle to Improve Treatment for Smokers in Public Housing
Brief Title: Intervention Study to Increase Smoking Cessation Rates Among Public Housing Residents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Harvard School of Public Health (HSPH) (Other); The Miriam Hospital (Other); Boston Housing Authority (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-28386; 1R01CA141587-03 (NIH)
Record Dates: First submitted 2012-07-24; First posted 2012-07-27 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2015-01

CONDITIONS: Tobacco Cessation
Keywords: Tobacco Cessation; Public Housing; Community Health Workers; Motivational Interviewing; Patient centered; Low-income; Tobacco Treatment Advocates; Social Epidemiology; Smoking cessation predictors; Behavioral Intervention; Non-pharmacologic
MeSH Terms: conditions — Tobacco Use Cessation | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Extensive TTA interaction (Experimental): Persons interested in quitting smoking will receive multiple in-person visits from a peer Tobacco Treatment Advocate (TTA) who will provide motivational interviewing, basic smoking cessation counseling assistance, navigation to smoking cessation resources, and social support.
  Interventions: Behavioral: Motivational interviewing; Behavioral: Smoking cessation counseling; Behavioral: Navigation to smoking cessation resources; Behavioral: Social support
- Minimal TTA interaction (Active Comparator): Persons interested in quitting smoking will receive a single in-person visit from a peer Tobacco Treatment Advocate (TTA) who will provide basic smoking cessation counseling assistance.
  Interventions: Behavioral: Smoking cessation counseling

INTERVENTIONS:
Behavioral: Motivational interviewing — The TTA will use motivational interviewing (MI) techniques to assess the participant's motivation and readiness to quit, suggest plans, and assist the participant in selecting a method of treatment.
  Arms: Extensive TTA interaction
Behavioral: Smoking cessation counseling — The TTA will provide information to the participant regarding evidence-based treatments for smoking cessation, including counseling and nicotine replacement therapy (NRT); assist in a quit plan; and discuss issues such as obtaining social support, staying in treatment, and dealing with lapses.
Behavioral: Navigation to smoking cessation resources — The TTA will assist participants in obtaining NRT and getting connected to smoking cessation counseling services, such as the Smokers' Quitline and clinic-based programs.
  Arms: Extensive TTA interaction
Behavioral: Social support — Meetings with the TTA will be a source of social support for the participant as they attempt to quit or stay quit.
  Arms: Extensive TTA interaction

SUMMARY:
The purpose of this study is to determine whether public housing residents trained in Tobacco Cessation and Motivational Interviewing Techniques to become Tobacco Treatment Advocates(TTA) will be effective in increasing the quit rate of smokers in Boston Public Housing. The investigators hypothesize that smokers that receive multiple TTA visits will be more likely to (1) use smoking cessation resources and (2) quit compared to smokers who receive a single visit.

DETAILED DESCRIPTION:
The study is a group-randomized trial in which 10 pubic housing developments (PHDs) are randomized to the experimental condition and 10 to the control condition. All smokers who enroll in the study at a particular PHD receive the same intervention. Smokers at control sites receive written materials that offer strategies for quitting and information about availability of treatment programs, as well as a one-time meeting with a Tobacco Treatment Advocate (TTA). The intervention group receives the same written materials but also has much more extensive interactions with a TTA. TTAs provide peer counseling (Peer Counseling is defined as: performance of limited counselor functions, under counselor supervision, by person of similar age,gender, race, ethnicity and/or SES of the counselee) to smokers during in- person Motivational Enhancement meetings (target range 7-9) as well as additional in person and phone contacts, as needed for each participant, over a 6-month period. TTAs receive intensive training in motivational interviewing and smoking cessation counseling deliver the intervention components (counseling activities and provision of environmental supports) in addition to encouraging utilization of smoking cessation treatment programs such as the Smokers' QuitLine (SQL) and clinic-based programs. In order to avoid the potential for contamination due to TTAs interacting with participants at both intervention and control sites, meetings with participants at control sites are conducted by special Control TTAs. Data are collected from study participants at baseline, 3 months, 7 months and 12 months, and also from the SQL and clinics.

ELIGIBILITY:
Inclusion Criteria:

* Current smoker, defined as having smoked in last 100days
* Housing Sites: Sites are eligible for the study if they have 50+ smokers determined by synthetic estimates based on citywide survey data.
* Age 18-79
* Current everyday or someday smokers
* Planning to quit smoking in 30 days or thinking about quitting in next 6 months,
* Have smoked 100 cigarettes in lifetime
* Speak English or Spanish
* Plan to live in Public Housing for next 12 months
* Able and willing to provide consent

Exclusion Criteria:

* Smokers less than 18 years of age at time of consent.
* Unable to communicate orally in English or Spanish.
* Currently using pharmacological treatment for smoking cessation
* Currently working with the Smokers Quitline or other Community Health Center based cessation program
* Cognitive/ psychiatric conditions that would interfere with ability to understand and participate in the study
* Have been abstinent for 7 or more days.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2011-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Point prevalence smoking abstinence | 7 months
  7 and 30-day abstinence from smoking by self-report with verification by carbon monoxide breath test

SECONDARY OUTCOMES:
Utilization of smoking cessation resources | 7 months
  Use of SQL, smoking cessation programs at health clinics or hospitals, physician counseling

OTHER OUTCOMES:
Medication use | 3 months, 7 months, 12 months
  Use of nicotine replacement therapy and/or other smoking cessation medications

CONTACTS AND LOCATIONS:
Overall Officials: Daniel R Brooks, DSc, Principal Investigator — Boston University
Locations (1):
- Boston University School of Public Health, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No